CLINICAL TRIAL: NCT02610985
Title: 3-dimensional Versus Conventional Laparoscopy in Patients Undergoing Total Hysterectomy for Benign Disease - A Randomised Clinical Trial
Brief Title: 2-D and 3-D Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Elise Hoffmann, MD, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2D/3D hysterectomy
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Fibroma, Bleeding
Keywords: Imaging, Three-Dimensional; Hysterectomy; laparoscopic hysterectomy
MeSH Terms: conditions — Fibroma; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2-Dimensional laparoscopic hysterectomy (Active Comparator): traditional 2-D laparoscopy
  Interventions: Device: 2-D laparoscopy
- 3-Dimensional laparoscopic hysterectomy (Experimental): experimental 3-D laparoscopy
  Interventions: Device: 3-D laparoscopy

INTERVENTIONS:
Device: 3-D laparoscopy — 3-D laparoscopy
  Arms: 3-Dimensional laparoscopic hysterectomy
Device: 2-D laparoscopy — 2-D laparoscopy
  Arms: 2-Dimensional laparoscopic hysterectomy

SUMMARY:
Background:

No randomised trials have been conducted, and only a single retrospective study exists comparing 3D and 2D laparoscopic hysterectomy. In that study, operative time for hysterectomy was significantly lower for 3D compared to 2D conventional laparoscopy. Complication rates were similar for the two groups. Thus, although one out of nine women is hysterectomized and although laparoscopy is one of the recommended routes of surgery, evidence whether to choose 2D laparoscopy, 3D laparoscopy is sparse.

Objective:

To compare pain and recurrence to usual activity level. Secondary to compare complications during the operation, postoperative complications, time to return to work, length of hospital stay and operative time.

Design:

Investigator-initiated, blinded, randomised controlled trial.

Intervention description:

Operative procedures follow the same principles and the same standard whether the surgeon's vision is 2D or 3D.

Trial size Roskilde/Herlev Hospital, Denmark:

200 patients in each arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for laparoscopic hysterectomy with or without bilateral salpingectomy or bilateral salpingooophorectomy for benign indications.

Exclusion Criteria:

* Women not suitable for laparoscopic hysterectomy including:

  * Ultrasound appraisal of uterus weight > 1000 gram
  * Need for prolapse surgery and therefore indication for vaginal hysterectomy.
* Inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Score on SF 36 psychical health survey 6 weeks after surgery | 6 weeks
Pain (VAS score) assessed immediately at return to the gynaecological unit (about 5 hours postoperatively) and (VAS score) in the morning days 1-3 postoperatively. | 3 days

SECONDARY OUTCOMES:
Major complications during the operation, postoperative complications | 6 weeks
Minor complications during the operation, postoperative complications | 6 weeks
Score on SF 36 mental health survey 6 weeks after surgery | 6 weeks
Length of hospital stay | 6 weeks
Operative time | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sjaellands Univercety Hospital, Roskilde, Region Sjælland, Denmark

REFERENCES:
- [Derived] Hoffmann E, Bennich G, Larsen CR, Lindschou J, Jakobsen JC, Lassen PD. 3-dimensional versus conventional laparoscopy for benign hysterectomy: protocol for a randomized clinical trial. BMC Womens Health. 2017 Sep 7;17(1):76. doi: 10.1186/s12905-017-0434-7. PMID 28882141